CLINICAL TRIAL: NCT06471582
Title: Implications for the Timing of Energy Availability on Menstrual Cycle Function
Brief Title: Timing of Energy Availability on Menstrual Cycle Function
Acronym: FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Colorado Springs (Other)
Responsible Party: Principal Investigator, Marissa Baranauskas, Assistant Professor, University of Colorado, Colorado Springs
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FAST
Record Dates: First submitted 2024-06-17; First posted 2024-06-24 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Menstrual Irregularity
Keywords: functional hypothalamic amenorrhea; menstrual cycle; female athlete
MeSH Terms: conditions — Menstruation Disturbances | interventions — Artificially Sweetened Beverages

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fed with Carbohydrates (Experimental): Participants will complete 3, 90-minute stationary cycle or treadmill exercise sessions 1 h after consuming a meal containing 1 g carbohydrate/ kg body weight. During exercise, they will consume an artificially sweetened beverage containing 0.7 g carbohydrate/ kg body mass/ h as a 2:1 mixture of glucose and fructose.
  Interventions: Dietary Supplement: Artificially Sweetened Carbohydrate Beverage
- Fasted without Carbohydrates (Placebo Comparator): Participants will complete 3, 90-minute stationary cycle or treadmill exercise sessions following an overnight fast. During exercise, they will consume an artificially sweetened beverage containing no carbohydrates.
  Interventions: Dietary Supplement: Artificially Sweetened Beverage

INTERVENTIONS:
Dietary Supplement: Artificially Sweetened Carbohydrate Beverage — Beverage containing 0.7 g carbohydrate/ kg body mass/ h as a 2:1 mixture of glucose and fructose and artificial sweetener
  Arms: Fed with Carbohydrates
Dietary Supplement: Artificially Sweetened Beverage — Beverage containing no carbohydrates or kilocalories and an artificial sweetener
  Arms: Fasted without Carbohydrates

SUMMARY:
The primary aim of this clinical trial is to evaluate how fasted prolonged exercise may influence circulating reproductive hormones (i.e., estradiol, progesterone, luteinizing hormone) and menstrual cycle length when energy availability is maintained at or above 30 kcal/kg lean body mass/ day among women who regularly do running or cycling exercise. A secondary aim is to determine the effects of fasted prolonged exercise on serum leptin and cortisol.

Participants will be asked to do the following over a ~3 month enrollment period:

* attend a laboratory visit at the beginning of the study to have their resting metabolic rate, aerobic fitness, and body composition tested
* monitor their menstrual cycle length, urine hormones, perceived stress levels, and diet for ~3 months
* complete 3, 90-minute exercise sessions on a stationary bike or treadmill either fed (consuming a carbohydrate meal 1 h prior and 0.7 g carbohydrate/ kg body mass/ h during exercise) or fasted (consuming no meal prior and no carbohydrates during exercise) during month ~3
* saliva samples will be taken prior to and after 90-minute exercise sessions for quantification of leptin and cortisol

ELIGIBILITY:
Inclusion Criteria:

* participates in structured running or cycling exercise for at least 30 minutes on 3 or more days per week
* accustomed to exercising for 90 minutes or more
* has regular periods every 21-35 days
* have not taken hormonal contraceptives for at least the past 6 months
* is not currently or trying to become pregnant or breastfeeding, and has not been pregnant or breastfeeding in the past 12 months
* does not currently have a diagnosis of a major menstrual cycle disorder (i.e., amenorrhea, polycystic ovary syndrome [PCOS], endometriosis, ovarian cancer, ovarian insufficiency, uterine or endometrial cancer)
* does not currently have a metabolic disease (i.e., hypothyroidism, hyperthyroidism, Cushing disease, Addison's disease, diabetes, congenital adrenal hyperplasia)
* does not currently have a major cardiovascular or respiratory disease

Exclusion Criteria:

* miss more than 7 consecutive days of aerobic activity (i.e., running, cycling, cross training)
* demonstrate clinical low energy availability as defined as energy availability <30 kcal/kg fat free mass
* report menstrual cycle lengths <21 or >35 days in the first 2 months of at-home monitoring
* do not demonstrate an anticipated rise in luteinizing hormone and progesterone in the first 2 months of at-home monitoring
* begin taking a hormonal contraceptive
* become pregnant
* are diagnosed with a menstrual cycle disorder (i.e., amenorrhea, polycystic ovary syndrome [PCOS], endometriosis, ovarian cancer, ovarian insufficiency, uterine, or endometrial cancer)
* are diagnosed with a metabolic disease (i.e., hypothyroidism, hyperthyroidism, Cushing disease, Addison's disease, diabetes)
* are diagnosed with a major cardiovascular or respiratory disease
* are unable to follow instructions for any of the procedures

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Urinary estrone-3-glucuronide (E3G) | 3 months
  ng/mL
Urinary pregnanediol glucuronide (PdG) | 3 months
  ug/mL
Urinary luteinizing hormone (LH) | 3 months
  MIU/mL
Menstrual cycle length | 3 months
  days

SECONDARY OUTCOMES:
Salivary cortisol | 3 days
  ng/mL
Salivary leptin | 3 days
  ng/mL

CONTACTS AND LOCATIONS:
Locations (1):
- William J. Hybl Sports Medicine and Performance Center, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No